CLINICAL TRIAL: NCT02145806
Title: Validation of Korean Version of ICIQ-SF
Status: Completed | Type: Observational
Sponsor: The Catholic University of Korea (Other)
Collaborators: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Yeon Hee Kim, Assistant professor, The Catholic University of Korea
Other Study IDs: CMC_UI_2014
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Urinary Incontinence
Keywords: Urinary incontinence; Validation study; Pregnant women; Postpartum period
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No

SUMMARY:
1. Validation of the Korean version of the ICIQ-UI SF for pregnant and postpartum women
2. Evaluation the effect of urinary incontinence in pregnant and postpartum women.

ELIGIBILITY:
Inclusion Criteria:

* Being pregnant or postpartum ≤ 3 weeks
* Able to read and understand Korean
* At least 18 years of age

Exclusion Criteria:

* Refuse to participate in the study
* Pelvic inflammatory disease
* Psychiatric disease
* Needed to be treated in the 7 days

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 130
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Urinary incontinence | 1-2 weeks